CLINICAL TRIAL: NCT07350408
Title: Mapping Post-falls Management Organisational Processes for Older People Who Fall in Care Homes in England
Brief Title: Mapping Post-falls Organisational Processes in Care Homes
Acronym: Post-falls
Status: Recruiting | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 25HC001
Record Dates: First submitted 2025-12-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-11

CONDITIONS: Fall
Keywords: falls; implementation science; care homes; long-term care; organisational management

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to map post-falls management organisational processes for older people in care homes. The main question to answer is 'What post-falls management organisational processes are used for older people in care homes?' Participants (care home and healthcare staff) will complete a one off online national survey about policies and processes relating to falls management in their organisation.

ELIGIBILITY:
Inclusion Criteria:

* Care home staff in any role or healthcare staff in any role working in a primary, community, emergency and acute settings
* Work in a care home or healthcare setting in England
* Has any previous experience in supporting older people immediately after a fall in a care home as part of their role
* Aged 16 years or over

Exclusion Criteria:

* Care home and healthcare staff working outside of England
* Staff working outside of stated settings
* No experience in supporting older people immediately after a fall in a care home as part of their role
* Under 16 years of age

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Care home staff in any role or healthcare staff in any role working in a primary, community, emergency and acute settings in England, with experience of supporting older people immediately after a fall in a care home as part of their role
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
post-falls practices for older people in care homes | Baseline only
  The survey collects information about current policies and procedures being used to manage falls in care homes. This is a one off cross-sectional survey to collect this information at a single time point.

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham University Hospital NHS Trust, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The anonymised Excel file containing survey responses will be made available upon request, for supporting further research and ensuring transparency, by contacting the CI after the results have been published. Sharing the file will require sponsor approval. The file will not contain identifiable information. The spreadsheet will be sent securely from an NHS.net email address. There will be no geographical restrictions. Sharing research data will be in line with the NIHR's commitment to open access of research outputs
Time Frame: After publication
Access Criteria: For research purposes Sponsor approval required No geographical restrictions